CLINICAL TRIAL: NCT04760795
Title: Stress, Personality, Attachment and Coping During the Covid Crisis.
Acronym: STERACOVID
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN922020
Record Dates: First submitted 2021-02-17; First posted 2021-02-18 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Psychiatric Disorder; Aging
Keywords: COVID-19; teleconsultation; Stress; containment; post-traumatic stress
MeSH Terms: conditions — Mental Disorders; COVID-19 | interventions — Weights and Measures; Patient Health Questionnaire

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- coping strategy based on problem: 59 geriatric patients will be included on the group: coping strategy based on problem
  Interventions: Other: PTSD Check List (PCL) scale; Other: Brief COPE scale; Other: GAD-7 (Generalized Anxiety Disorder) scale (during containment); Other: Analog scale; Other: GAD-7 (Generalized Anxiety Disorder) scale (post containment); Other: Big Five Inventory (BFI) scale; Other: Relationship Scales Questionnaire (RSQ)
- coping strategy based on emotion: 59 geriatric patients will be included on the group: coping strategy based on emotion
  Interventions: Other: PTSD Check List (PCL) scale; Other: Brief COPE scale; Other: GAD-7 (Generalized Anxiety Disorder) scale (during containment); Other: Analog scale; Other: GAD-7 (Generalized Anxiety Disorder) scale (post containment); Other: Big Five Inventory (BFI) scale; Other: Relationship Scales Questionnaire (RSQ)

INTERVENTIONS:
Other: PTSD Check List (PCL) scale — PTSD Check List (PCL) scale will be realized to evaluated post-traumatic stress disorder.
Other: Brief COPE scale — Brief COPE scale dispositional version will be realized to evaluated usual coping strategies. It was assessed during the teleconsultations and post containment.
Other: GAD-7 (Generalized Anxiety Disorder) scale (during containment) — GAD 7 (Generalized Anxiety Disorder) scale will be realized to evaluated anxiety during containment. It was assessed during the teleconsultations.
Other: Analog scale — Analog scale will be realized to evaluated anxiety during containment. It was assessed during the teleconsultations.
Other: GAD-7 (Generalized Anxiety Disorder) scale (post containment) — GAD-7 (Generalized Anxiety Disorder) scale will be realized to evaluated anxiety during post containment.
Other: Big Five Inventory (BFI) scale — Big Five Inventory (BFI) will be realized to evaluated personality.
Other: Relationship Scales Questionnaire (RSQ) — Relationship Scales Questionnaire (RSQ) will be realized to evaluated attachment style.

SUMMARY:
Because of containment due to Covid-19, the French High Authority for Health (HAS) recommended reinforced monitoring of patients taken in care in the psychiatric ward, with special attention for people over the age of 65. To meet this recommendation, the geriatrics department of the hospital of Charity of Saint-Etienne hospital and the Vinatier hospital in Lyon organized follow-up of these patients by telephone throughout the containment period, thus allowing continuity of care. This pandemic situation and these measures are unprecedented; it is difficult to anticipate the psychological impact on patients.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate if the type of coping strategies usually employed has an effect on the outbreak of a post-traumatic stress after containment. In addition, a second part of the study will propose to assess the factors influencing the experience of containment such as personality, attachment style or coping strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients followed by teleconsultation during containment due to COVID 19
* Patient affiliated or entitled to a social security scheme
* Patient who received informed information about the study and who co-signed, with the investigator, a consent to participate in the study (for the part excluding routine care).

Exclusion Criteria:

- Major neurocognitive disorder

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged of 65 years old et taken in care in the psychiatric ward will be included.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2022-10-19 (Actual)

PRIMARY OUTCOMES:
Analysis post traumatic stress disorder measured by PTSD Check List (PCL) results | Year: 1
  The PTSD Check List (PCL) is a self-questionnaire to assess the post traumatic stress disorder and contains 17 items with minimum score 17 (no post traumatic stress disorder) and maximum score at 85 (post traumatic stress disorder important).

SECONDARY OUTCOMES:
Analysis usual coping strategies measured by brief COPE (dispositional version) results | Year: 1
  Brief COPE (dispositional version) is a questionnaire to assess the usual coping strategies and contains 28 items with minimum score 28 (not at all) and maximum score at 112 (a lot).
Analysis of situation of patients | Year: 1
  It is composite of analysis of socio-demographic data, conditions of confinement, diagnostic elements. It was collected in the medical record.
Analysis usual coping strategies during containment measured by brief COPE (dispositional version) results | Year: 1
  Brief COPE (dispositional version) is a questionnaire to assess the usual coping strategies during containment and contains 28 items with minimum score 28 (not at all) and maximum score at 112 (a lot).
Analysis anxiety during containment measured by GAD-7 (Generalized Anxiety Disorder) results | Year: 1
  GAD-7 (Generalized Anxiety Disorder) is a questionnaire to assess the anxiety during containment and contains 7 items with minimum score 0 (not anxiety) and maximum score at 21 (anxiety).
Analysis anxiety related to the containment context measured by analogue scale | Year: 1
  Analogue scale contains minimum score 0 (absence of stress) and maximum score at 10 (stress maximal).
Analysis anxiety post containment measured by GAD-7 (Generalized Anxiety Disorder) results | Year: 1
  GAD-7 (Generalized Anxiety Disorder) is a questionnaire to assess the anxiety post containment and contains 7 items with minimum score 0 (not anxiety) and maximum score at 21 (anxiety).
Analysis of personalities by Big Five Inventory (BFI) scale | Year: 1
  Big Five Inventory (BFI) scale to assess the personalities and contains 45 items with 5 dimensions: openness, awareness, extroversion, agreeableness and neurosis.
Analysis attachment measured by Relationship Scales Questionnaire (RSQ) scale results | Year: 1
  Relationship Scales Questionnaire (RSQ) scale is a questionnaire to assess attachment style and contains 30 items to identify 2 latent dimensions: the "model of oneself" and the "model of the others".
presence of traumatic life events | Year: 1
  Analysis of presence of traumatic life events

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Rouch, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (2):
- France (2):
  - CH Le Vinatier, Bron
  - Chu Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pongan E, Rouch I, Herrmann M, Perrot C, Lebrun-Givois C, Spirli L, Briollet C, Martin HS, Laurent B, Bachelet R, El Haouari H, Buisson A, Edjolo A, Dorey JM. Anxiety symptoms during COVID-19 in older adults with psychiatric disorders. Front Psychiatry. 2023 Jan 16;13:1082807. doi: 10.3389/fpsyt.2022.1082807. eCollection 2022. PMID 36741567
- [Derived] Edjolo A, Dorey JM, Herrmann M, Perrot C, Lebrun-Givois C, Buisson A, El Haouari H, Laurent B, Pongan E, Rouch I. Stress, Personality, Attachment, and Coping Strategies During the COVID-19 Pandemic: The STERACOVID Prospective Cohort Study Protocol. Front Psychiatry. 2022 Jun 27;13:918428. doi: 10.3389/fpsyt.2022.918428. eCollection 2022. PMID 35832598